CLINICAL TRIAL: NCT02240654
Title: Evaluation of Potential Off-label Use of Dabigatran Etexilate in Europe
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.144
Record Dates: First submitted 2014-09-15; First posted 2014-09-16 (Estimated); Results first posted 2017-10-16 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Dabigatran etexilate

SUMMARY:
This is a descriptive, observational, multi-country European cross-sectional study of new users of dabigatran etexilate that aims to characterise on- and off-label status and other medical characteristics at the time of the first captured prescription of dabigatran etexilate in each database. The study will be conducted using Cegedim Strategic Database (CSD, France), Danish National Databases (Denmark) and Clinical Practice Research Datalink (CPRD, UK).

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Have at least 1 year of enrolment in the electronic database.
2. Have not been prescribed dabigatran etexilate during the 1-year period prior to the index date.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New users of dabigatran etexilate in each database
Sampling Method: Non-Probability Sample
Enrollment: 36573 (Actual)
Dates: Start 2014-11-28 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1160.144.1 Boehringer Ingelheim Investigational Site, Barcelona, Spain

REFERENCES:
- [Derived] Cainzos-Achirica M, Varas-Lorenzo C, Pottegard A, Asmar J, Plana E, Rasmussen L, Bizouard G, Forns J, Hellfritzsch M, Zint K, Perez-Gutthann S, Pladevall-Vila M. Methodological challenges when evaluating potential off-label prescribing of drugs using electronic health care databases: A case study of dabigatran etexilate in Europe. Pharmacoepidemiol Drug Saf. 2018 Jul;27(7):713-723. doi: 10.1002/pds.4416. Epub 2018 Mar 23. PMID 29570897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a descriptive, observational, non-interventional (NIS) multinational, European cross-sectional study with sources of information for clinical conditions available being highly variable across countries/data sources
Pre-assignment Details: Because it is not possible to rule out duplicate patients across the 2 French panels, all numbers were calculated stratified by data source, and for France further stratified by panel - i.e., not overall.
Groups:
- Dabigatran Etexilate (Pradaxa®)_France (Cardiologists): New users of Dabigatran etexilate (Pradaxa capsules, 75 mg, 110 mg and 150 mg) identified from panels of cardiologists in Cegedim Strategic Data Longitudinal Patient Database (CSD-LPD) in France (primary care information)
- Dabigatran Etexilate (Pradaxa®)_France (GPs): New users of Dabigatran etexilate (Pradaxa capsules, 75 mg, 110 mg and 150 mg) identified from panels of general practitioners (GPs) in Cegedim Strategic Data Longitudinal Patient Database (CSD-LPD) in France (primary care information)
- Dabigatran Etexilate (Pradaxa®)_Denmark: New users of Dabigatran etexilate (Pradaxa capsules, 75 mg, 110 mg and 150 mg) in National Health Databases in Denmark (DK) (hospital episodes, dispensed ambulatory medications)
- Dabigatran Etexilate (Pradaxa®)_UK (HES Linkable): New users of Dabigatran etexilate (Pradaxa capsules, 75 mg, 110 mg and 150 mg) in Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK) Hospital Episode Statistics (HES) linkable (primary care information, hospital episodes, dispensed ambulatory medications)
- Dabigatran Etexilate (Pradaxa®)_UK (HES Non-linkable): New users of Dabigatran etexilate (Pradaxa capsules, 75 mg, 110 mg and 150 mg) in Clinical Practice Research Datalink (CPRD) in the United Kingdom (UK) non-linkable HES (primary care information)
Period: Overall Study
Arm/Group | Dabigatran Etexilate (Pradaxa®)_France (Cardiologists) | Dabigatran Etexilate (Pradaxa®)_France (GPs) | Dabigatran Etexilate (Pradaxa®)_Denmark | Dabigatran Etexilate (Pradaxa®)_UK (HES Linkable) | Dabigatran Etexilate (Pradaxa®)_UK (HES Non-linkable)
Started | 1706 | 2813 | 28619 | 2150 | 1285
Completed | 1706 | 2813 | 28619 | 2150 | 1285
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study population included new users of dabigatran etexilate in the study period. New users were defined as those patients who initiated treatment with dabigatran etexilate during the study period and who had not used it during the previous year.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabigatran Etexilate (Pradaxa®)_France (Cardiologists) | Dabigatran Etexilate (Pradaxa®)_France (GPs) | Dabigatran Etexilate (Pradaxa®)_Denmark | Dabigatran Etexilate (Pradaxa®)_UK (HES Linkable) | Dabigatran Etexilate (Pradaxa®)_UK (HES Non-linkable) | Total
Number analyzed (Participants) | 1706 | 2813 | 28619 | 2150 | 1285 | 36573
Age, Continuous [Mean (Standard Deviation); unit: years] — Because it is not possible to rule out duplicate patients across the 2 French panels, all numbers were calculated stratified by data source, and for France further stratified by panel - i.e., not overall. Totals computed here may not be correct, as those assume that there were no duplicate patients in CSD-LPD.
  years | 75.5 (10.0) | 74.0 (10.4) | 71.8 (10.9) | 74.1 (11.2) | 73.1 (11.5) | NA (NA) — Because it is not possible to rule out duplicate patients across the 2 French panels, all numbers were calculated stratified by data source, and for France further stratified by panel - i.e., not overall.
Sex: Female, Male [Count of Participants; unit: Participants] — For 282 patients, information on gender was missing. Because it is not possible to rule out duplicate patients across the 2 French panels, all numbers were calculated stratified by data source, and for France further stratified by panel - i.e., not overall.
  Total (men, women) may not be correct, as those assume that there were no duplicate patients in CSD-LPD.
  Participants
    Female | NA — 599 female patients and gender for 282 patients was missing | 1272 | 13567 | 938 | 571 | NA — Total not calculated because data are not available (NA) in one or more arms.
    Male | NA — 825 patients and gender for 282 patients was missing | 1541 | 15052 | 1212 | 714 | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Potential Off-label Use Estimated Among New Users of Dabigatran Etexilate in Each of the Data Sources.
Description: Definition of off-label use of oral dabigatran etexilate (DE) was based on use for a disease/medical condition other than labelled indications,as described/documented in the data source used in the respective countries, taking into account the changes in the label within the study period. The prevalence of potential off-label use among new users of DE during the overall study period is calculated as the proportion of patients meeting the definition of off-label use by dividing the number of index prescriptions that represented off-label use by the total number of index prescriptions.
  Two definitions were applied to estimate potential off-label use based on either recorded diagnoses or proxies: a broad definition of on-label prescribing using codes for disease indication e.g.atrial fibrillation(AF) and a restrictive definition excluding patients with conditions for which the drug is not indicated e.g.valvular AF.
  SPAF:Stroke & systemic embolism in adult patients with non-valvular AF
Time Frame: Time period since approval of the SPAF indication in, France: 01 August 2011 to 30 June 2014; Denmark: 01 August 2011 to 30 November 2013; UK: 01 August 2011 to 30 August 2015.
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dabigatran Etexilate (Pradaxa®)_France (Cardiologists) | Dabigatran Etexilate (Pradaxa®)_France (GPs) | Dabigatran Etexilate (Pradaxa®)_Denmark | Dabigatran Etexilate (Pradaxa®)_UK (HES Linkable) | Dabigatran Etexilate (Pradaxa®)_UK (HES Non-linkable)
Number analyzed (Participants) | 1706 | 2813 | 28619 | 2150 | 1285
percentage of participants
  Broad definition | 24.1 [22.1 to 26.1] | 34.0 [32.3 to 35.8] | 17.1 [16.6 to 17.5] | 5.7 [4.7 to 6.7] | 11.5 [9.8 to 13.4]
  Restrictive definition | 37.5 [35.2 to 39.8] | 44.1 [42.2 to 45.9] | 29.1 [28.4 to 29.7] | 17.4 [15.8 to 19.1] | 25.6 [23.2 to 28.1]

ADVERSE EVENTS:
Description: International Society for Pharmacoepidemiology and European Medicines Agency guidelines state that NIS studies conducted using medical chart reviews/electronic claims/health care records do not require expedited reporting of suspected Adverse events (AEs)/reactions.Given the type of data used for this study,no suspected AEs/reactions were reported
Arm/Group | Dabigatran Etexilate (Pradaxa®)_France (Cardiologists) | Dabigatran Etexilate (Pradaxa®)_France (GPs) | Dabigatran Etexilate (Pradaxa®)_Denmark | Dabigatran Etexilate (Pradaxa®)_UK (HES Linkable) | Dabigatran Etexilate (Pradaxa®)_UK (HES Non-linkable)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Clinical information being highly variable across countries was likely to be major driver of different proportions.UK(HES link) is likely to provide most accurate estimate(France and DK data need to be interpreted cautiously because of limited info)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.